CLINICAL TRIAL: NCT06373250
Title: Maternal Consequences of Membrane Stripping During Vaginal Birth
Brief Title: Maternal Consequences of Membrane Stripping
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Sena Dilek Aksoy, Principal Investigator, Kocaeli University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: sdilek7
Record Dates: First submitted 2024-04-13; First posted 2024-04-18 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-04

CONDITIONS: Maternal Care for Other Abnormalities of Cervix
Keywords: stripping; vaginal birth; pain; cervix; membrane
MeSH Terms: conditions — Pain | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Membrane stripping group (Active Comparator): Participants in the membrane stripping group will be stripped at least once during labour. A visual analog scale will be completed before and after each vaginal examination. During the vaginal examination, the Bishop scoring form will be filled out. The average of the visual analogue scale and Bishop scores obtained during the vaginal examinations is taken. Bleeding will be assessed by weighing the pads at four hours postpartum. You will also be asked to complete the short form of the Birth Satisfaction Scale.
  Interventions: Behavioral: Membrane stripping group
- Control group (Active Comparator): Participants in the control group will not undergo any membrane stripping or other cervical interventions during labour, and other routine procedures will be carried out. A visual analog scale will be completed before and after each vaginal examination. During the vaginal examination, the Bishop scoring form will be filled out. The average of the visual analogue scale and Bishop scores obtained during the vaginal examinations is taken. Bleeding will be assessed by weighing the pads at four hours postpartum. You will also be asked to complete the short form of the Birth Satisfaction Scale.
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Membrane stripping group — An information form will be filled in for admission to the Primipar participating maternity unit. Membrane stripping will be performed during a vaginal examination at least once during the birth process. A visual analog scale will be completed before and after each vaginal examination. During the vaginal examination, the Bishop scoring form will be filled out. The average of the visual analogue scale and Bishop scores obtained during the vaginal examinations will be taken. At four hours postpartum, the pads are weighed and the amount of bleeding is recorded on the form. You will also be asked to complete the short form of the Birth Satisfaction Scale.
  Arms: Membrane stripping group
Other: Control group — You will be asked to fill in an information form to be admitted to the Primipar participating maternity unit. No membrane stripping are applied and no cervical interventions are made during the birth process. A visual analog scale will be completed before and after each vaginal examination. During the vaginal examination, the Bishop scoring form will be filled out. The average of the VAS and Bishop scores obtained during the vaginal examinations will be taken. At four hours postpartum, the pads are weighed and the amount of bleeding is recorded on the form. You will also be asked to complete the short form of the Birth Satisfaction Scale.
  Arms: Control group

SUMMARY:
This study aims to investigate the maternal effects of membrane stripping during vaginal birth. This study was designed as an experimental case-control study. The sample size in the study was determined by Njoku et al in 2023 to assess the effectiveness of membrane stripping applied to participants who had vaginal birth in reducing the incidence of prolonged pregnancy. Calculated based on the study conducted by. The sample size of the study was calculated using G*Power 3.1.9.2, and the mean and standard deviation of the Bishop score in the relevant article were used to calculate the effect size. Using the mean and standard deviation of the relevant article, the blended effect size was calculated as 0.596. The minimum number of individuals that should be included in the sample of this research was calculated using G*Power 3.1.9.2, effect size: 0.596, α= 0.05, power: 0.95 (stripping = 70, control = 70) and at least in each group in the sample size. The sample size was set at 70 participants. The research data will be collected by the researcher using the Informed Volunteer Consent Form, Participant Information Form, Bishop Scoring, Visual Analogue Scale, and Birth Satisfaction Scale Short Form, which were created by the researcher within the framework of the literature on the subject.

DETAILED DESCRIPTION:
Aim: This study was designed to investigate the maternal outcomes of membrane stripping during vaginal delivery.

H0: There is no difference between the maternal outcomes of pregnant women who underwent membrane stripping during vaginal delivery and those who did not.

H1: There is a difference in maternal outcomes between pregnant women who underwent membrane stripping during vaginal delivery and those who did not.

The research data will be collected by the researcher using the Informed Volunteer Consent Form, Participant Information Form, Bishop Scoring, Visual Analogue Scale and Birth Satisfaction Scale Short Form, which have been developed by the researcher from the literature on the subject.

Research application process After obtaining the necessary ethics committee and institutional permissions to conduct the research, the institution will be visited and participants who will give birth vaginally and meet the inclusion criteria for the research will be interviewed. Participants will be informed that they can participate in the study and leave the study at any time without affecting the care received in the hospital, and their voluntary consent will be obtained. Once participants are included in the study, they will be randomly assigned to membrane stripping and control groups. Membrane stripping will be applied at least once to the membrane stripping group, but will not be applied to the control group. Data will be collected through face-to-face interviews by researchers working in the hospital's delivery room. The Visual Analog Scale will be marked by the participants of the research. Visual analog scale will be filled in by case and control groups before and after routine vaginal examination. The Bishop Score will be completed during each vaginal examination. The average of the visual analog scale pain scores and Bishop scores obtained during vaginal examinations in the membrane stripping group and control group will be taken. The last bleeding control of both groups in the early postpartum period (the first 4 hours after birth) will be determined by weighing their pads and they will be asked to fill out the Birth Satisfaction Scale Short Form.

Data analysis Statistical analysis was performed using IBM SPSS Statistic 22.0 (IBM Corp., Armonk, NY, USA). Descriptive statistical methods (number, percentage, mean, standard deviation) will be used to evaluate socio-demographic data. If the data are found to be suitable for normal distribution, they will be analysed with parametric tests (Chi-square, T-test, etc.) in comparison with categorical variables, and if they are not found to be suitable for normal distribution, they will be analysed with non-parametric tests (Mann-Whitney U test, Kruskal Wallis, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Speak and understand Turkish,
* 18 years and older,
* In labour for vaginal birth,
* At term gestational age (37-41 weeks),
* Primiparous pregnant women,
* Not having a high-risk pregnancy,
* Head presentation,
* Without cephalopelvic disproportion,
* Have gone through active labour in hospital,
* Women who volunteer to take part in the research will be included.

Exclusion Criteria:

* Those who do not have sufficient mental health to fill out the survey form,
* Having a history of previous C/S,
* Caesarean section or interventional birth is planned,
* Intrauterine fetal ex,
* Pregnant women who wish to leave at any point in the study will be excluded.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 140 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale evaluation of vaginal examination pain | This scale will be filled in by the participants just before the vaginal examination.
  The patient marks his or her own pain on a 10 cm ruler, which says no pain on one end and the most severe pain on the other end. The patient is told that there are two endpoints and to mark anywhere between these points that matches the severity of the pain. The distance between the onset of no pain and this point marked by the patient is measured and recorded in centimeters. It is stated that visual analog scale is more sensitive and reliable than other unidimensional scales in pain severity measurement. The visual analog scale is more sensitive than the simple descriptive scale.
Visual analogue scale evaluation of vaginal examination pain | This scale will be filled in by the participants immediately after the vaginal examination.
  The patient marks his or her own pain on a 10 cm ruler, which says no pain on one end and the most severe pain on the other end. The patient is told that there are two endpoints and to mark anywhere between these points that matches the severity of the pain. The distance between the onset of no pain and this point marked by the patient is measured and recorded in centimeters. It is stated that visual analog scale is more sensitive and reliable than other unidimensional scales in pain severity measurement. The visual analog scale is more sensitive than the simple descriptive scale.
Evaluation of the cervix with Bishop score | This scale will be evaluated by the researcher during the vaginal examination at the beginning of labor.
  Bishop score is used to evaluate dilation, effacement, level, consistency and position of the cervix.
Evaluation of the amount of bleeding | The amount of bleeding will be determined by weighing all pads used in the first 4 hours after birth.
  During the early postpartum period, the amount of bleeding will be determined by weighing the participant's pads.
Birth Satisfaction Scale Short Form | The participant will be asked to fill it in at the fourth hour after birth.
  The Birth Satisfaction Scale-Short Form is a 10-item Likert scale. It consists of 3 sub-dimensions: quality of care, personal characteristics of the woman and stress experienced during childbirth. The lowest score on the scale is "0" and the highest score is "40", and as the score on the scale increases, so does the level of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Sena Dilek Aksoy, Ph.D., Principal Investigator — Kocaeli University; Burcu Ozturk, M.Sc., Study Chair — Duzce Ataturk State Hospital; Beyza Akbaba, Study Chair — Duzce Ataturk State Hospital
Locations (1):
- Kocaeli University, Köseköy, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salau JO, Onile TG, Musa AO, Gbejegbe EH, Adewole AA, Olorunfemi GO, Olumodeji AM. Effectiveness and safety of membrane sweeping in the prevention of post-term pregnancy: a randomised controlled trial. J Obstet Gynaecol. 2022 Oct;42(7):3026-3032. doi: 10.1080/01443615.2022.2126752. Epub 2022 Sep 30. PMID 36178679